CLINICAL TRIAL: NCT05004064
Title: Phase II Study of Acalabrutinib and Rituximab for Elderly or Frail Patients With Previously Untreated Mantle Cell Lymphoma
Brief Title: Acalabrutinib and Rituximab in Previously Untreated Mantle Cell Lymphoma
Acronym: CARAMEL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCL/137775; 2021-002393-42 (EudraCT Number)
Record Dates: First submitted 2021-06-08; First posted 2021-08-13 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2024-10

CONDITIONS: Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — acalabrutinib; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Acalabrutinib and rituximab (Experimental): Patients with untreated mantle cell lymphoma will receive acalabrutinib and rituximab for up to six cycles. Each cycle will comprise of acalabrutinib 100mg twice daily orally for 28 days and rituximab 375mg/m2 IV on day 1 (+/1 3 days) of every cycle.
  Interventions: Drug: Acalabrutinib; Drug: Rituximab

INTERVENTIONS:
Drug: Acalabrutinib — Patients will receive acalabrutinib 100mg twice daily for up to six 28 day cycles. Patients can receive 100mg once daily for cycle 1, day 1 to day 7, according to the investigator's discretion.
Drug: Rituximab — Patient will receive rituximab 375 mg/m2 IV on day 1 (+/- 3 days) of each cycle, for a maximum of 6 cycles

SUMMARY:
This is a phase II, single-arm, open-label, multicentre study of acalabrutinib and rituximab for elderly or frail patients with previously untreated mantle cell lymphoma.

DETAILED DESCRIPTION:
This is a Phase II, multicentre, single arm, open label pilot study to assess the safety and efficacy of acalabrutinib in combination with rituximab for previously untreated elderly frail mantle cell lymphoma patients.

48 patients will be recruited from 12 UK centres over 30 months.

Patients will receive acalabrutinib and rituximab for up to six cycles. The cycle length is 28 days. Specifically, patients will receive acalabrutinib, orally, at a dose of 100 mg twice daily for 28 days and rituximab 375 mg/m2 intravenously on day 1 (+/-3) of each cycle.* Patients with any degree of response at the Week 12 (end of cycle 3) and Week 24 assessments (end of cycle 6) will continue with acalabrutinib monotherapy at a dose of 100 mg twice daily until disease progression, the development of unacceptable toxicity or any other reason (whichever occurs sooner).

* Note: Acalabrutinib may be administered at a dose of 100 mg od po for cycle 1 day 1-7 at the local investigator's discretion. The dose should be escalated to full dose (100 mg bd) by day 8, cycle 1 if no toxicity is seen (see dose modification section). If a patient experiences toxicity during cycle 1 day 1-7 100 mg od po, the case must be discussed with the TMG to decide if acalabrutinib should continue. The CTC CARAMEL team should be contacted as soon as possible to arrange discussions with the TMG. Rituximab may be administered subcutaneously at a flat dose of 1400 mg from cycle 2 onwards following an intravenous dose of 375 mg/m2 in cycle 1. Consider splitting the first dose of rituximab at cycle 1 in the minority of MCL patients presenting with a white cell count of >25 x 109/L. Consider splitting 25-50 mg/m2 on D1 and 325-350 mg/m2 on D2 of cycle 1 (to a total of 375 mg/m2 over D1/D2) according to investigator and site preference. Full dose 375 mg/m2 IV (or s/c equivalent) should be given in all patients from cycle 2 as a single dose.

All patients will be followed up for a minimum of 2 years following being registered into the trial. For patients that have been in follow-up for more than 2 years, annual survival and disease status follow-up will continue until the end of the trial.

ELIGIBILITY:
Inclusion criteria:

1. Men and women ≥ 60 years of age.
2. Pathologically confirmed MCL, with documentation of monoclonal B cells that have a chromosome translocation t(11;14)(q13;q32) and/or overexpress cyclin D1.
3. Stage II-IV MCL and requiring treatment in the opinion of the treating clinician.
4. Eastern Cooperative Oncology Group (ECOG) performance status 0-3
5. One or more of the following:

   * Age 80 years or more
   * Cumulative Illness Rating Scale for Geriatrics (CIRS-G) score 6 or greater
   * Left ventricular ejection fraction (LVEF) less than or equal to 50% as assessed by echocardiogram
   * Significant co-morbidities or cardiac risk factors making anthracycline-containing chemotherapy inadvisable
   * Heart failure clinically determined by the presence of New York Heart Association (NYHA) failure grade II due to a cause other than MCL
   * Impaired respiratory function with DLCO and/or FVC/FEV1 ratio less than 75% of predicted due to a cause other than MCL
   * Significant respiratory illness e.g. moderate chronic obstructive pulmonary disease (COPD) bronchiectasis
   * Other co-morbidities that in the Investigator's opinion which would preclude the use of standard full dose immuno-chemotherapy (to be discussed on a case-by-case basis with the TMG, via UCL CTC)
6. Willing and able to participate in all required evaluations and procedures in this study protocol including swallowing capsules/tablets without difficulty.
7. Negative serum or urine pregnancy test for women of childbearing potential (WOCBP).
8. Willing to comply with the contraceptive requirements of the trial.
9. Written informed consent.

Exclusion criteria:

1. Any prior therapy (including targeted inhibitors) for MCL (other than prior localised radiotherapy, a 10-day pulse of high dose steroids or continuous prednisolone above 20mg od or equivalent for symptom control).
2. Patients considered by the investigator fit enough to receive standard, full dose cytotoxic immunochemotherapy as treatment for non-transplant eligible MCL e.g., full dose R-CHOP, VR-CAP, R-Bendamustine, R-FC.
3. Prior malignancy (or any other malignancy requiring active treatment), except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, localised prostate cancer or other cancer from which the subject has been disease free for ≥ 2 years or which will not limit survival to < 5 years.
4. Clinically significant cardiovascular disease such as uncontrolled arrhythmias, or myocardial infarction within 6 months of screening, or any Class 3 or 4 cardiac disease as defined by the New York Heart Association (NYHA) Functional Classification (33), or corrected QT interval (QTc) > 480 msec at screening.
5. Malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel that is likely to affect absorption, symptomatic inflammatory bowel disease, partial or complete bowel obstruction, or gastric restrictions and bariatric surgery, such as gastric bypass.
6. Known history of infection with HIV or any uncontrolled active systemic infection (e.g., bacterial, viral or fungal).
7. Known history of drug-specific hypersensitivity or anaphylaxis to any study drug (including active product or excipient components).
8. Active bleeding or history of bleeding diathesis (e.g. haemophilia or von Willebrand disease).
9. Uncontrolled AIHA (autoimmune haemolytic anaemia) or ITP (idiopathic thrombocytopenic purpura).
10. Known presence of a gastrointestinal ulcer diagnosed by endoscopy within 3 months before screening.
11. Requires treatment with a strong cytochrome P450 3A4 (CYP3A4) inhibitor/inducer.
12. Requires or receiving anticoagulation with warfarin or equivalent vitamin K antagonists (e.g. phenprocoumon) within 7 days prior to the first dose of study drug.
13. Prothrombin time (PT)/INR or aPTT (in the absence of lupus anticoagulant) > 2 x upper limit of normal (ULN).
14. Requires treatment with proton pump inhibitors (e.g. omeprazole, esomeprazole, lansoprazole, rabeprazole, or pantoprazole). Subjects receiving proton pump inhibitors who switch to H2-receptor antagonists or antacids are eligible for enrolment to this study.
15. History of significant cerebrovascular disease/event, including stroke or intracranial haemorrhage, within 6 months before the first dose of study drug.
16. Major surgical procedure within 28 days prior to the first dose of study drug. Note: If a subject had major surgery, they must have recovered adequately from any toxicity and/or complications from the intervention before the first dose of study drug.
17. Hepatitis B or C serologic status: subjects who are hepatitis B core antibody (anti-HB core) positive and who are surface antigen negative will need to have a negative polymerase chain reaction (PCR) test. Those who are hepatitis B surface antigen (HbsAg) positive or hepatitis B PCR positive will be excluded. Those who are hepatitis C antibody or PCR positive will be excluded (those who are hepatitis C antibody positive but PCR negative will not be excluded). Note, if a patient with known HBV or HCV infection who is on current antiviral treatment meets serology criteria for trial eligibility then the case must be discussed with the TMG prior to registering the patient.
18. Absolute neutrophil count <1.0 x 109/L (or requires growth factor support to maintain absolute neutrophil count >1.0 x 109/L) and/or platelets <75 x109/L unless related to bone marrow infiltration or splenomegaly due to underlying MCL (where platelets between 50-75 x109/L are acceptable)
19. Total bilirubin > 1.5 x ULN, unless due to Gilbert's syndrome or of non-hepatic origin.
20. AST and/or ALT > 3 x ULN.
21. Calculated creatinine clearance <30 mL/min.
22. History of or ongoing confirmed central nervous system (CNS) involvement
23. Breastfeeding or pregnant.
24. Concurrent participation in another therapeutic clinical trial.
25. Live vaccine within 28 days prior to the first study drug dose

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-11-30 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | 24 weeks
  To determine the efficacy of acalabrutinib in combination with rituximab in terms of disease response.

SECONDARY OUTCOMES:
Progression free survival | From the date of first dose of acalabrutinib until the date of progression or death. Assessed up to 42 months.
  Progression free survival measured from the date of first dose of acalabrutinib until the date of first documented progression or date of death from any cause.
Overall survival | From the date of first dose of acalabrutinib until the date of death. Assessed up to 42 months.
  Overall survival measured from the date of first dose of acalabrutinib until the date of death from any cause.
Quality of life up to 24 months | At baseline, week 12, week 24, month 12 and month 24
  The EORTC QLQ-C30 will be used to measure participant-assessed quality of life
Incidence and frequency of grade 1-2 and 3+ adverse events seen in both treatment arms. | Between the start of study treatment and 30 calendar days post last IMP administration.
  Safety and toxicity will be characterised in terms of adverse events as assessed by CTCAE v5.0. The incidence and frequency of adverse events during treatment and after treatment will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Toby Eyre, Principal Investigator — Churchill Hospital, Oxford, United Kingdom
Locations (12):
- United Kingdom (12):
  - The Royal Bournemouth Hospital, Bournemouth
  - University Hospital of Wales, Cardiff
  - Royal Cornwall Hospital, Cornwall
  - Beatson West of Scotland Cancer Centre, Glasgow
  - St. Bartholomew's Hospital, London
  - University College London Hospital, London
  - The Christie Hospital, Manchester
  - Clatterbridge Cancer Centre, Metropolitan Borough of Wirral
  - Norfolk and Norwich University Hospital, Norwich
  - Cancer and Haematology Centre, Churchill Hospital, Oxford
  - Derriford Hospital, Plymouth
  - Royal Stoke Hospital, Stoke-on-Trent

IPD SHARING:
Plan to Share IPD: No